CLINICAL TRIAL: NCT03125616
Title: Babies Born Early Antibody Response to Men B Vaccination: A Phase IV Multicentre Randomised Study to Evaluate the Primary and Booster Immune Responses in UK Preterm Infants Receiving Routine Immunisations and Incorporating a Three Dose Versus a Two Dose Schedule of 4CMenB (Bexsero®) for Primary Immunisation.
Brief Title: Babies Born Early Antibody Response to Men B Vaccination: BEAR Men B
Acronym: BEAR Men B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: GlaxoSmithKline (Industry); MeningitisNow (Unknown); Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16.0247; 2017-001487-38 (EudraCT Number)
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Prematurity; Vaccination; Meningococcal Disease
Keywords: Prematurity; Vaccination
MeSH Terms: conditions — Premature Birth; Meningococcal Infections | interventions — 4CMenB vaccine

STUDY DESIGN:
Intervention Model Description: This will be an open label, phase IV study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard UK 4CMenB vaccine (Active Comparator): 4CMenB (Bexsero®) vaccination at 2 and 4 months and a booster at 12 months .
  Interventions: Biological: 4CMenB Vaccine
- Additional 4CMenB Vaccine (Experimental): 4CMenB (Bexsero®) vaccination at 2, 3 and 4 months and a booster at 12 months.
  Interventions: Biological: 4CMenB Vaccine

INTERVENTIONS:
Biological: 4CMenB Vaccine — The infants will receive an intramuscular injection of the 4CMenB vaccine at 2 months
  Other Names: Bexsero
Biological: 4CMenB Vaccine — The infants will receive an intramuscular injection of the 4CMenB vaccine at 3 months
  Other Names: Bexsero
  Arms: Additional 4CMenB Vaccine
Biological: 4CMenB Vaccine — The infants will receive an intramuscular injection of the 4CMenB vaccine at 4 months
  Other Names: Bexsero
Biological: 4CMenB Vaccine — The infants will receive an intramuscular injection of the 4CMenB vaccine at 12 months
  Other Names: Bexsero

SUMMARY:
In the UK, babies receive their vaccinations according to a standard schedule, irrespective of their gestation at birth. This policy is designed so that all babies are protected as early as possible from vaccine preventable diseases such as polio, diphtheria, tetanus, rotavirus, pertussis (whooping cough), Haemophilus influenzae type B, pneumococcal disease and now meningococcal B disease. The 4CMenB vaccination (Bexsero®) was added to the UK schedule in September 2015 and there has been no research looking at whether the vaccine gives the same protection to babies born early as it does to those born at term. The Investigators want to compare two different schedules of 4CMenB and see if one gives better protection to babies born prematurely. It is possible that an extra 4CMenB dose (i.e. three doses in early infancy instead of two) will offer better protection for premature babies. This is what the Investigators are trying to find out through this study.

DETAILED DESCRIPTION:
This will be an open label, phase IV study. After appropriate consent, 132 premature infants born at <35 weeks gestation (i.e. up to 34 weeks and 6 days), 50% <30 weeks gestation (i.e. up to 29 weeks and 6 days) will be randomised to 1 of 2 4CMen B schedules either at 2,4 and 12 months or 2,3,4 and 12 months. Babies will remain in the study for around 12 months, from recruitment to 13 months of age. All visits can be performed at the participant's home or in clinic, depending on the preference of the parents and study team.

Blood samples will be obtained at 5 months of age (post primary sample), 12 months (persistence sample) and 13 months (post booster sample). Reactogenicity and safety will be assessed by caregiver completion of a 7-day diary after each vaccine dose. Inpatients will be monitored for cardiorespiratory events for 72 hours after vaccination by healthcare staff and this information will be collected on the CRF. This will include details of oxygen saturations, heart rate, respiratory rate and details of any episodes of desaturation, bradycardia or apnoea. Particular emphasis will be placed on rates, timing and intensity of fever and other adverse reactions in the first 24 hours after vaccination, because this remains a cause of great concern amongst neonatologists.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant born at <35 weeks gestation
* No contraindications to vaccination according to the 'Green Book'
* Willing and able to comply with study procedures
* Written informed consent

Exclusion Criteria:

* Contraindication to vaccination according to the Green Book
* Life-limiting congenital abnormality or condition
* Prior diagnosis of an immunodeficiency syndrome
* Considered unlikely to complete expected follow up until the end of the study

Ages: 7 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
hSBA GMT | Tested in each infant at 5 months of age (1 month after completion of primary vaccinations)
  hSBA GMT one month after completing primary immunisations for relevant 4CMenB (Bexsero®) antigens: fHbp, NadA and PorA
hSBA proportions | Tested in each infant at 5 months of age (1 month after completion of primary vaccinations)
  hSBA proportions ≥ 1:4, one month after completing primary immunisations for relevant 4CMenB (Bexsero®) antigens: fHbp, NadA and PorA.

SECONDARY OUTCOMES:
Reactions within 7 days | Assessed in each infant for the 7 days following vaccination
  The percentage of infants experiencing fever, local reactions and non-febrile systemic reactions within the 7 days following each vaccine dose
Cardiorespiratory status for 72 hours following vaccination | Assessed in all infants in hospital for 72 hours following vaccination
  The percentage of inpatients experiencing change / deterioration in cardiorespiratory status within the 72 hours following each vaccine dose
Suspicion of sepsis in 7 days following vaccination | Assessed in all infants in the 7 days following vaccination
  The percentage of infants investigated for sepsis and commenced on antibiotics within 7 days of vaccination
Fever and/or suspicion of sepsis in the 28 days following vaccination | Assessed in all infants in the 28 days following vaccination
  The percentage of infants who experience fever and/or are investigated for sepsis and commenced on antibiotics within 28 days of vaccination
Serious adverse events | Assessed in all infants at the conclusion of the study
  The percentage of infants who experience a serious adverse event at any point within the study
Persistence of hSBA GMTs | Assessed in all infants at 12 months of age
  hSBA GMTs at 12 months of age (pre booster) for relevant 4CMenB (Bexsero®) antigens: fHbp, NadA and PorA
Persistence of hSBA proportions ≥1:4 | Assessed in all infants at 12 months of age
  hSBA proportions ≥1:4, at 12 months of age (pre booster) for relevant 4CMenB (Bexsero®) antigens: fHbp, NadA and PorA
Booster response: hSBA GMTs | Assessed in all infants at 13 months of age
  hSBA GMTs at 13 months of age (post booster) for relevant 4CMenB (Bexsero®) antigens: fHbp, NadA and PorA;
Booster response: hSBA proportions ≥1:4 | Assessed in all infants at 13 months of age
  hSBA proportions ≥1:4, at 13 months of age (post booster) for relevant 4CMenB (Bexsero®) antigens: fHbp, NadA and PorA.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Heath, MBBS, Principal Investigator — St George's, University of London
Locations (1):
- St Georges University Hospital NHS Foundation Trust, Tooting, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Derived] Daniel O, Srikanth S, Clarke P, Le Doare K, Heath PT, Jones CE, Scorrer T, Snape M, Calvert A. Pertussis antibody responses in infants born to mothers vaccinated at different time points in pregnancy. Vaccine. 2025 Aug 30;62:127481. doi: 10.1016/j.vaccine.2025.127481. Epub 2025 Jul 12. PMID 40652683
- [Derived] Calvert A, Andrews N, Barlow S, Borrow R, Black C, Bromage B, Carr J, Clarke P, Collinson AC, Few K, Hayward N, Jones CE, Le Doare K, Ladhani SN, Louth J, Papadopoulou G, Pople M, Scorrer T, Snape MD, Heath PT. An open-label, phase IV randomised controlled trial of two schedules of a four-component meningococcal B vaccine in UK preterm infants. Arch Dis Child. 2024 Oct 18;109(11):898-904. doi: 10.1136/archdischild-2024-327040. PMID 38977298
- See also: Meningococcal: the green book, chapter 22 — https://www.gov.uk/government/publications/meningococcal-the-green-book-chapter-22